CLINICAL TRIAL: NCT05165160
Title: Local Undertaking of Resected Non-small Cell Lung Cancer by Generating a Residual Disease Outline Based on Circulating Cell-free DNA
Brief Title: Residual Disease Evaluation of Resected NSCLC by cirDNA Analysis
Acronym: LUNGDOC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL20_0548
Record Dates: First submitted 2021-12-17; First posted 2021-12-21 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Nsclc
Keywords: Stage I to IIIA; Performance status 0-2; Written and signed informed consent form
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eligible patients (Experimental)
  Interventions: Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: Blood sample — Pre- and postoperative blood sample

SUMMARY:
Prognosis of resectable early stages NSCLC might be improved by a better knowledge of post-operative minimal residual disease (MRD). This could be achieved by studying patient with stage I to IIIA completely resected-NSCLC, comparing qualitative and quantitative features of pre- and post-operative circulating cell-free DNA (cirDNA), using MiTest. We assume that the evolution of the parameters of MiTest and relapse rate after surgery are related and expect to prove that normalization of MiTest at one month after surgery is a prognostic factor of reduced relapse at one year.

DETAILED DESCRIPTION:
Rationale: Non-small cell lung cancer (NSCLC) is the most lethal cancer worldwide with an increasing incidence each year and a better prognosis for resectable early stages, despite frequent recurrences. Yet, oncologic adjuvant cares are decided without accurate information about minimal residual disease (MRD).

The improvement of post-operative management of early-stage NSCLC supposes to better understand post-operative MRD. In a cancer screening study performed recently, we showed that nuclear and mitochondrial circulating cell-free DNA (cirDNA) are significantly modified in cancer situation and might stand as promising surrogates of MRD. The analysis of cirDNA in blood with quantitative PCR (qPCR), through the use of multi-analyte test called MiTest, could offer a very sensitive study model of MRD in patients with resected NSCLC. We assume that the evolution of these parameters and relapse rate after surgery are related and expect to prove that normalization of MiTest at one month after surgery is a prognostic factor of reduced relapse at one year.

Main objective: Our main objective is to determine whether the lack of normalization of MiTest of cirDNA one month after the resection of an early-stage NSCLC is predictive of relapse rate at 1 year.

Methodology: The RD-CD LUNGDOC Project is a monocentric, prospective, interventional, non-comparative, single-arm prognostic exploratory study in which we estimated 120 patients as the number of subjects needed. Subjects will be included consecutively at the Montpellier Academic Hospital and blood sampled at 3 timepoints: once before surgery and twice after surgery, at one month and one year.

Main inclusion criteria: patients with resected NSCLC, stage I to IIIA, performance status 0-2, normal end organ functions.

Main non-inclusion criteria: previous systemic neoadjuvant treatment, resection margins R1 and R2, neoadjuvant treatment received, non-invasive lung carcinoma, multiple primary lung cancer, previous malignancy during the past 3 years, concomitant primitive malignant disease.

Primary endpoint: Recurrence- free survival (RFS) probability according to MiTest at 1 year after surgery.

Secondary endpoints: Overall survival (OS) probability according to MiTest at one month and at one-year post-surgery, qualitative and quantitative features of cirDNA.

Feasibility: CirDNA analysis will be performed at the Montpellier Cancer Research Institute in the of Alain THIERRY's team "Biomarkers in precision oncology team".

Expected results and prospects: We expect to prove that normalization of MiTest at one month after surgery is a prognostic factor for patients with resected NSCLC, which could deeply modify management of resected NSCLC by better stratifying prognosis and possibly anticipating relapses.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or older
* Patients with a resectable NSCLC
* Definite stage I to IIIA
* Performance status of 0, 1 or 2
* Normal end organ functions
* Written and signed informed consent form
* Subjects must be covered by public health insurance.

Exclusion Criteria:

* Any previous systemic neoadjuvant treatment: targeted therapy, chemotherapy, immune checkpoint blockade
* Previous radiotherapeutic neoadjuvant treatment
* Resection margins R1 and R2
* Non-invasive lung carcinoma
* Multiple primary lung cancer.
* Previous malignancy during the past 3 years (except non-melanomatous skin cancer)
* Preexisting interstitial lung disease
* known HIV, active viral B hepatitis or C hepatitis
* Patient with any other situation responsible for cirDNA rate increasing (active auto-immune disease, 10 days following blood transfusion)
* Patient unable to attend all scheduled visits
* Woman of childbearing age without efficient contraception, breastfeeding
* Patient with a legal protection measure (guardianship, curatorship)
* Vulnerable patient protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival probability according to MiTest at one year after surgery (RFS1) | The year after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Montpellier, France